CLINICAL TRIAL: NCT01393522
Title: A Randomized Double Blind Placebo Control Trial of Milnacipran for Migraine Pain
Brief Title: Study Evaluated the Effectiveness of Milnacipran to Reduce Pain Levels in Individuals With Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Smith (Other)
Responsible Party: Sponsor-Investigator, Timothy Smith, Vice President of Clinical Research, St. John's Mercy Research Institute, St. Louis
Organization: Mercy Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SAV-MD-25
Record Dates: First submitted 2011-07-06; First posted 2011-07-13 (Estimated); Results first posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Chronic Migraine
Keywords: headache; migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Milnacipran; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milnacipran (Active Comparator): Oral Milnacipran titration was Day 1-2 - 12.5mg/d; Day 3-6 - 12.5mg bid; Day 7-14 - 25mg bid; Day 15 and on - 50mg bid. After the first 30 days, patients did not continue to increase the dose beyond the dose they have achieved at 30 days. At study completion medication taper as follows: patients who at their completion visit were taking 50mg bid decreased to 25mg bid for 4 days, then decreased to 12.5mg bid for 2 days, then 12.5mg once a day for one day and then stopped. Patients on 25mg bid, decreased to 12.5mg bid for 2 days, 12.5mg once a day for one day and then stopped.
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator): Sugar Pill No active ingredients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — titration schedule starting with 12.5mg per day increasing to 50mg twice a day, starting with day 1 to day 90 and then taper down as appropriate for dose.
  Other Names: Savella
  Arms: Milnacipran
Drug: Placebo — Placebo dosing schedule was Day 1-2, 1 tablet daily, Day 3-6 BID, Day 7-14 BID, Day 15 an on through day 90 BID and taper down
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if milnacipran taken twice daily is effective in reduction of headache pain.

DETAILED DESCRIPTION:
Milnacipran is a serotonin norepinephrine reubtake inhibitor (SNRI) approved for the management of fibromyalgia in the United States.

Migraine and fibromyalgia have significant co-morbidity. Of 100 patients with fibromyalgia, 76% had chronic headaches, of whom 63% had migraine. Interestingly, general measures of pain, disability, sleep quality, and psychological distress were similar in individuals with fibromyalgia with and without headache. Conversely, the prevalence of fibromyalgia in women with migraine was reported as 22%, and at a headache referral center, 36% of headache patients had fibromyalgia.

Because of significant co-morbidity, as well as the likelihood of shared pathophysiologic mechanisms, there is reason to believe that a medication effective for fibromyalgia might reduce migraine pain, especially where the pain has taken on the nature of a chronic pain disorder, as in chronic migraine. The current study evaluated the benefits of milnacipran in individuals with chronic migraine.

Patients with chronic migraine were randomized to either Milnacipran or Placebo. Patients completed 30 days of baseline followed by 90 days of headache diaries while taking assigned medication. Primary outcomes were reduction in pain severity and improvement in migraine specific quality of life (MSQ) while secondary outcomes included reduction in migraine and non-migraine headache days and symptomatic use of medication for migraine. Independent sample t-tests were used to evaluate the changes in primary and secondary measures between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the age of 18 and 65
* Headache fulfills ICHD-2 criteria for: chronic migraine, or probable medication overuse headache where individual headaches meet criteria for migraine
* At least 15 headache days/month and at least 8 migraine or probable migraine days/month for the past 3 months, by patient report (including days of headache relieved with a triptan or related compound).
* Age at onset of chronic migraine < 60 years old

Exclusion Criteria:

* Pregnancy or attempting conception
* Unable to read or write English
* Use of Opiates >/= 10 days per month
* Subject has failed >/= 4 adequate preventive trials of antidepressant medications due to lack of efficacy; at least one trial included another SNRI.(An adequate preventive trial defined as at least 6 weeks on therapeutic dose [150mg of amitriptyline or nortriptyline or other tricyclic, 150mg of venlafaxine, 60mg of duloxetine])
* Subjects on antidepressant medications, including SNRIs who cannot safely withdraw from those medications, in the assessment of the PI. Subjects on other headache preventives (beta blockers, antiepileptic drugs), at stable dose for at least three months, will be allowed to participate.

A. Subjects on other headache preventives may be included in the study if the medication has been at a stable dose for 3 months.

* Presence of fibromyalgia or another pain or medical disorder that would make it difficult for patient to distinguish headache-related quality of life from overall health related quality of life.
* Uncontrolled or unstable psychiatric disorder (PHQ-9 score or GAD-7 score >15 with sentinel questions >/=4, or in opinion of examiner), or anticipated need for change in psychotropic medications during duration of study period; or suicidality.
* Chronic kidney disease, liver disease, or any poorly controlled medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Smith, MD, Principal Investigator — Mercy Research
Locations (2):
- United States (2):
  - Mercy Health Research, St Louis, Missouri
  - Headache Wellness Center, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from two Headache focused ambulatory clinics. From Q2, 2011 until Q2, 2013. Recruitment involved printed flyers placed in the examination rooms of both sites as well as clinical staff informing patients about the study opportunity.
Pre-assignment Details: Patients completed a 30 day run-in period prior to randomization to ensure that they were accurate and compliant in completing diaries and experiencing sufficient headaches. Specifically they were required to have > 15 headache days and 8 (probable) migraine days . Patients below this threshold but met other headache criteria could be eligible.
Groups:
- Milnacipran: Milnacipran: titration schedule starting with 12.5mg per day increasing to 50mg twice a day, starting with day 1 to day 90 and then will taper down.
- Placebo: Placebo: Tablet will be titrated 1 tablet once a day increased per protocol to 2 tablets twice a day, with a starting dose of 12.5mg per day to 50 mg twice a day
Period: Overall Study
Arm/Group | Milnacipran | Placebo
Started | 19 | 18
Completed | 12 | 14
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milnacipran | Placebo | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.63 (9.59) | 37.39 (15.07) | 38.01 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian_Non Hispanic | 17 | 15 | 32
  Non_Caucasian | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 37
Years with Headache [Mean (Standard Deviation); unit: years] | 20.44 (13.51) | 17.89 (9.69) | 19.20 (11.65)
Pain Severity [Mean (Standard Deviation); unit: units on a scale] — On headache days, patients were instructed to complete a Visual Analog Scale (VAS) to rate their pain intensity. Their response (the scale was 100 cm long) was measured and assigned a score (0-100) with higher numbers indicating more severity.
  units on a scale | 57.67 (11.60) | 61.87 (17.95) | 59.71 (14.69)
MIgraine Days Per Month [Mean (Standard Deviation); unit: Number of Days with Migraine per Month] — On days where the patient indicated they had a headache, patients were instructed to complete the diary questions with headache characteristics (using International Headache Classification criteria). This information was used to calculate migraine days per month.
  Number of Days with Migraine per Month | 10.72 (6.79) | 11.26 (5.35) | 10.98 (6.09)
MSQ- Preventive [Mean (Standard Deviation); unit: Standard Score] — Migraine Specific Quality of Life - Preventive. The Migraine Specific Quality of Life measures the impact Migraine has on the patient's Quality of Life. The Preventive subscale assesses the extent to which migraine prevents the patient's function. The subscale is measured on a standard scale from 0-100, where higher scores indicate better quality of life.
  Standard Score | 53.89 (21.04) | 47.78 (22.83) | 50.92 (21.91)
MSQ- Restrictive [Mean (Standard Deviation); unit: Standard Score] — Migraine Specific Quality of Life - Restrictive. The Migraine Specific Quality of Life measures the impact Migraine has on the patient's Quality of Life. The Restrictive subscale assesses the extent to which migraine restricts the patient's function. The subscale is measured on a standard scale from 0-100, where higher scores indicate better quality of life.
  Standard Score | 37.78 (13.63) | 33.68 (18.58) | 35.79 (16.04)
MSQ-Emotional [Mean (Standard Deviation); unit: Standard Score] — Migraine Specific Quality of Life - Emotional. The Migraine Specific Quality of Life measures the impact Migraine has on the patient's Quality of Life. The Emotional subscale assesses the extent to which migraine influences the patient's emotional function. The subscale is measured on a standard scale from 0-100, where higher scores indicate better quality of life.
  Standard Score | 38.15 (20.43) | 30.53 (26.14) | 34.44 (23.21)
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire - 9
  PHQ-9 total score ranges from 0 to 27. The Patient Health Questionnaire assesses depression symptoms. The higher the score, the more symptoms of depression and more severe the depression.
  PHQ-9 score total of 0-4 points equals minimal depression, 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
  units on a scale | 3.78 (3.12) | 5.05 (4.18) | 4.40 (3.64)
GAD-7 [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder - 7
  GAD-7 total score ranges from 0 to 21. The higher the score, the more symptoms of anxiety and more severe the anxiety.
  0-4 points equals minimal anxiety, 5-9 points indicates mild anxiety, 10-14 points indicates moderate anxiety, 15-21 points indicate severe anxiety.
  units on a scale | 2.89 (3.63) | 3.74 (3.94) | 3.30 (3.78)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 29.67 (7.62) | 28.32 (5.93) | 29.01 (6.80)
Blood Pressure - Systolic [Mean (Standard Deviation); unit: mmHg] | 120.83 (13.43) | 114.47 (13.34) | 117.74 (13.39)
Blood Pressure - Diastolic [Mean (Standard Deviation); unit: mmHg] | 74.67 (11.66) | 76.83 (8.84) | 75.72 (10.29)
Pulse [Mean (Standard Deviation); unit: Beats Per Minute] | 74.44 (8.26) | 75.47 (9.62) | 74.94 (10.61)
Non-Migraine Headache Days [Mean (Standard Deviation); unit: Days w/ Non-Migraine Headache per Month] — On days where the patient indicated they had a headache, patients were instructed to complete the diary questions with headache characteristics (using International Headache Classification criteria). This information was used to calculate non-migraine days per month.
  Days w/ Non-Migraine Headache per Month | 11.41 (8.02) | 10.65 (5.80) | 11.04 (6.94)
Days Using Medication for Headache Per Month [Mean (Standard Deviation); unit: Days per Month] — Patients indicated whether they took an acute medication for the treatment of headache that day. This information was used to calculate medication days per month.
  Days per Month | 15.59 (3.22) | 14.63 (7.22) | 15.12 (5.17)

OUTCOME MEASURES:

1. Primary Outcome: Change in VAS Pain Severity
Description: On headache days, patients were instructed to complete a Visual Analog Scale (VAS) to rate their pain intensity. Their response (the scale was 100 cm long) was measured and assigned a score (0-100) with higher numbers indicating more severity. Scores were averaged over a 30 day period to create the score for a time period (baseline and 90 days). Change in Pain score = Score[Baseline] - Score[90 days]. Higher scores indicate greater pain reduction.
Time Frame: Baseline and 90 days
Population: Intent to treat population (all participants who were randomized to one of the conditions and treated at least one migraine with Milnacipran or Placebo).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 3.23 [2.10 to 4.37] | 5.36 [4.25 to 6.45]
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.1, ANCOVA
Statistical Analysis 2: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.88, t-test, 2 sided

2. Secondary Outcome: Change in Days With Migraine Per Month From Baseline to 90 Days
Description: On days where the patient indicated they had a headache, patients were instructed to complete the diary questions regarding headache characteristics using International Headache Classification Diagnostics. This information was used to calculate migraine days per month. Days with migraine over a 30 day period were summed to generate a number for each time frame (baseline and 90 days). For the outcome measure, higher positive numbers indicate higher reduction of days with migraine.
  Change in days with migraine = Score[Baseline] - Score[90days]
Time Frame: Baseline and 90 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days per Month
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 19 | 18
Days per Month | 3.34 [3.13 to 3.54] | 4.62 [4.42 to 4.84]
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.33, t-test, 2 sided

3. Primary Outcome: Change in Migraine Specific Quality of Life - Restrictive
Description: The Migraine Specific Quality of Life measures the impact Migraine has on the patient's Quality of Life. The Restrictive subscale assesses the extent to which migraine restricts the patient's function. The subscale is measured on a standard scale from 0-100, where higher scores indicate better quality of life. For the outcome assessing change, higher positive scores indicate better outcomes.
Time Frame: Baseline and 90 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 21.01 [17.31 to 24.72] | 35.03 [31.43 to 38.62]
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.75, ANCOVA
Statistical Analysis 2: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.24, t-test, 2 sided

4. Primary Outcome: Change in Migraine Specific Quality of Life - Preventive
Description: The Migraine Specific Quality of Life measures the impact Migraine has on the patient's Quality of Life. The Preventive subscale assesses the extent to which migraine prevents the patient's function. The subscale is measured on a standard scale from 0-100, where higher scores indicate better quality of life. For the outcome assessing change, higher positive scores indicate better outcomes.
Time Frame: Baseline and 90 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 21.61 [21.46 to 21.77] | 31.26 [31.10 to 31.42]
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.16, t-test, 2 sided

5. Primary Outcome: Change in Migraine Specific Quality of Life - Emotional
Description: The Migraine Specific Quality of Life measures the impact Migraine has on the patient's Quality of Life. The Emotional subscale assesses the extent to which migraine influences the patient's emotional function. The subscale is measured on a standard scale from 0-100, where higher scores indicate better quality of life. For the outcome assessing change, higher positive scores indicate better outcomes.
Time Frame: Baseline and 90 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 29.89 [28.68 to 31.12] | 37.99 [36.81 to 39.18]
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.41, t-test, 2 sided

6. Secondary Outcome: Change in Days With Non-Migraine Headache Per Month From Baseline to 90 Days
Description: On days where the patient indicated they had a headache, patients were instructed to complete the diary questions regarding headache characteristics using International Headache Classification Diagnostics. This was information was used to calculate non-migraine headache days days per month. Days with migraine over a 30 day period were summed to generate a number for each time frame (baseline and 90 days). For the outcome measure, higher positive numbers indicate higher reduction of days with non-migraine headache.
  Change in days with non-migraine headache = Score[Baseline] - Score[90 days]
Time Frame: Baseline and 90 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days per Month
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 19 | 18
Days per Month | 2.35 [1.81 to 2.89] | 0.76 [0.22 to 1.31]
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.09, t-test, 2 sided

7. Secondary Outcome: Change in Days Using Headache Medication Per Month From Baseline to 90 Days
Description: On days where the patient indicated they had a headache (i.e., migraine or non-migraine headache), patients were instructed to complete the diary questions regarding whether they used medication to treat headache pain and related symptoms. This was used to calculate days using headache medication days per month. Days with migraine over a 30 day period were summed to generate a number for each time frame (baseline and 90 days). For the outcome measure, higher positive numbers indicate higher reduction of days using headache medication per month.
  Change in days using headache medication = Score[Baseline] - Score[90 days]
Time Frame: Baseline and 90 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days per Month
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 19 | 18
Days per Month | 1.28 [-0.17 to 2.75] | 2.17 [0.79 to 3.54]
Statistical Analysis 1: Comparison: Milnacipran vs Placebo; Test type: Superiority or Other; p = 0.78, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Milnacipran | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 5/19 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=19) | Placebo (N=18)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
testicular discomfort (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Given that the number needed to have adequate power to demonstrate differences was 38.3% higher than the number enrolled, it is difficult to make any specific conclusions about the efficacy of Milnacipran.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No